CLINICAL TRIAL: NCT02215174
Title: Rosuvastatin Pharmacokinetic (PK) Study in Caucasian and Asian Morbid Obese Patients
Brief Title: Rosuvastatin Interethnic PK Study
Acronym: RST
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: IRB approval expired
Sponsor: University of California, San Francisco (Other)
Collaborators: E-DA Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 14-13695.; 14-13695 (Other: University of California, San Francisco)
Record Dates: First submitted 2014-07-31; First posted 2014-08-13 (Estimated); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Statin Pharmacokinetics Pre and Post Gastric Bypass Surgery
Keywords: Rosuvastatin; PK; Interethnic; Morbid obese
MeSH Terms: interventions — Rosuvastatin Calcium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Asians (Experimental): Drug: Rosuvastatin Rosuvastatin 20mg po x1 Other Name: Crestor
  Interventions: Drug: Rosuvastatin
- Caucasians (Experimental): Drug: Rosuvastatin Rosuvastatin 20mg po x1 Other Name: Crestor
  Interventions: Drug: Rosuvastatin

INTERVENTIONS:
Drug: Rosuvastatin — Rosuvastatin 20mg po x1
  Other Names: Crestor

SUMMARY:
Statins are the first-line and most commonly prescribed drugs for the prevention of cardiovascular diseases and stroke in the world. Our preliminary studies suggest that Caucasians might have a higher risk of developing potentially life-threatening drug-drug interactions than Asians when taking statins. Drug-drug interactions occur in the body when two or more drugs interact in a way that alters their effectiveness and/or toxicity. These interactions are becoming an increasingly severe problem with statin usage since patients at higher risk for cardiovascular diseases also take statins combined with many other drugs, such as antihypertensive and diabetic drugs. Our study is aimed at understanding the molecular factors and providing a sound basis for the interethnic dosage and response differences for statins.

Drug-transporting proteins in intestine and liver tissues are responsible for taking up statins into the blood. It is hypothesized that there are interethnic function differences of these proteins and that they account for differences in statin blood levels between Caucasians and Asians and the frequency and/or severity of their respective drug-drug interactions. A clinical study will be conducted with Caucasian and Asian subjects undergoing gastric bypass surgery so excess intestine and liver tissue can be acquired as part of the standard procedure. Protein levels will be quantified in the tissues and correlate them with different statin blood levels.

ELIGIBILITY:
Inclusion Criteria:

* Subjects that are scheduled for bariatric surgery.
* Subjects that are able and willing to donate surplus intestinal tissue.
* Subjects with solute carrier organic anion transporter *1 (SLCO1B1) and breast cancer resistant protein (BCRP) 421CC genotypes.
* White/Caucasian/European and Asian/East Asian heritage individuals, male or female, 18 years of age or older.
* BMI between 30-55 kg/m2
* Be able to read, speak, and understand English(UCSF) and Chinese(Taiwan).
* Subjects capable of providing informed consent and completing the requirements of the study.

Exclusion Criteria:

* Subjects with active liver and kidney problems, severe cardiovascular diseases, type I diabetes, advanced pulmonary disease, and cancers.
* Subjects on chronic prescription or over the counter medication that have previously been reported to exhibit drug-drug interactions with rosuvastatin and cannot be stopped two weeks prior to and during the study, including gemfibrozil, cyclosporine, atazanavir, lopinavir and ritonavir.
* Subjects incapable of multiple blood draws (HCT < 30mg/dL).
* Subjects with a history of rhabdomyolysis.
* Subjects with a history of drug-related myalgias.
* Subjects with a history or diagnosis of hemorrhagic tendencies or blood dyscrasias.
* Subjects with a history of GI bleed or peptic ulcer disease.
* Subjects with a recent history of trauma.
* Subjects who smoke tobacco or have ongoing alcohol or illegal drug use.
* Subjects who are pregnant, lactating, or trying to conceive during the study period.
* Subjects allergic to rosuvastatin or any known component of the medications.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2015-02; Primary Completion 2018-12-06 (Actual); Study Completion 2018-12-06 (Actual)

PRIMARY OUTCOMES:
Area-under-the-concentration curve (AUC) of rosuvastatin | 0,1,2,3,4,5,6,8,12,24,36,48 hr post dosing

SECONDARY OUTCOMES:
Change in oral clearance of rosuvastatin | Pre-surgery period: 48 hr after dosing; post-surgery period: 48 hr after dosing. Two periods separated by at least two months.
  Changes in oral clearance of rosuvastatin within gastric bypass surgery will be analyzed using the ratio of areas under the systemic concentration curves (AUCs) from before to after surgery using the bioequivalence criteria of 80-125%. The oral clearance will be calculated based on the plasma data from each of the blood draws after the dosing period is completed (48hr). The pre and post surgery period are separated by at least a 8-week recovery period.
Descriptive comparison of messenger ribonucleic acid (mRNA) and protein expression in the tissues | Day of the surgery
  Tissue samples will be collected on the day of the surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Leslie Benet, PhD, Principal Investigator — University of California, San Francisco
Locations (2):
- University of California, San Francisco, San Francisco, California, United States
- E-Da Hospital, Kaohsiung City, Taiwan

REFERENCES:
- [Derived] Wu HF, Hristeva N, Chang J, Liang X, Li R, Frassetto L, Benet LZ. Rosuvastatin Pharmacokinetics in Asian and White Subjects Wild Type for Both OATP1B1 and BCRP Under Control and Inhibited Conditions. J Pharm Sci. 2017 Sep;106(9):2751-2757. doi: 10.1016/j.xphs.2017.03.027. Epub 2017 Apr 3. PMID 28385543